CLINICAL TRIAL: NCT01711970
Title: A Phase I/II Trial of Multiple Dose VB-111 and Weekly Paclitaxel for the Treatment of Recurrent Platinum-Resistant Müllerian Cancer
Brief Title: A Phase I/II Trial of VB-111 and Paclitaxel for Recurrent Platinum-Resistant Müllerian Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Vascular Biogenics Ltd. operating as VBL Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VB-111-157; 11-418 (Other: DF/HCC); NCT01801215 (obsolete NCT alias)
Record Dates: First submitted 2012-10-18; First posted 2012-10-23 (Estimated); Last update posted 2020-04-24 (Actual); Status verified 2020-04

CONDITIONS: Platinum Resistant Ovarian Cancer
MeSH Terms: interventions — Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- VB-111 (Experimental)
  Interventions: Drug: Paclitaxel

INTERVENTIONS:
Drug: Paclitaxel

SUMMARY:
This is a prospective, open label, dose escalating, Phase I/II study, measuring mainly the safety and tolerability of the combination of intravenous administration of VB-111 and paclitaxel in patients with platinum resistant ovarian cancer.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged > 18
* Histologically confirmed epithelial ovarian, peritoneal, or fallopian tube cancer, and uterine papillary serous carcinomas (UPSC), and gynecologic malignant mixed müllerian tumors (MMMTs).
* Must have had prior platinum or platinum based therapy.
* Eastern Cooperative Oncology Group (ECOG) status 0-1.
* Platinum resistant or refractory disease within 6 months of completing or while receiving a platinum and taxane containing regimen
* Measurable disease
* Adequate bone marrow and hematological function.
* Must have recovered from acute toxicity from prior treatment
* Prior treatment with an anti-angiogenic agent is not an exclusion criterion.
* No prior GI perforation, or GI obstruction or involvement of the bowel on imaging
* Known hypersensitivity to Cremophor EL. However, participants are eligible if they have had a prior paclitaxel reaction, but subsequently tolerated the drug at rechallenge.
* No patients receiving other investigational therapy for the past 30 days before dosing.

Exclusion Criteria:

* More than 3 prior lines of chemotherapy for recurrent cancer.
* History of other active malignancy, other than superficial basal cell and superficial squamous cell, or carcinoma in situ of the cervix within last 2 years.
* Life expectancy of less than 3 months
* CTC Grade 1 or greater neuropathy (motor or sensory) from comorbidity other than prior taxane exposure, such as diabetes.
* Inadequately controlled hypertension or prior history of hypertensive crisis or hypertensive encephalopathy.
* New York Heart Association (NYHA) Grade II or greater congestive heart failure.
* History of myocardial infarction or unstable angina within 6 months prior to study Day 1.
* History of stroke or transient ischemic attack within 6 months prior to Day 1.
* Known CNS disease, except for treated brain metastasis
* Significant vascular disease (e.g., aortic aneurysm, requiring surgical repair or recent peripheral arterial thrombosis) within 6 months prior to Day 1.
* History of hemoptysis (1/2 teaspoon of bright red blood per episode) within 1 month prior to Day 1.
* Evidence of bleeding diathesis or significant coagulopathy (in the absence of therapeutic anticoagulation).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Estimated)
Dates: Start 2012-11; Primary Completion 2017-05-03 (Actual); Study Completion 2017-05-03 (Actual)

PRIMARY OUTCOMES:
Define toxicities | 2 years
  Define toxicities of a limited number of doses of combination VB-111 and weekly paclitaxel spanning anticipated effective doses.

CONTACTS AND LOCATIONS:
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Arend RC, Beer HM, Cohen YC, Berlin S, Birrer MJ, Campos SM, Rachmilewitz Minei T, Harats D, Wall JA, Foxall ME, Penson RT. Ofranergene obadenovec (VB-111) in platinum-resistant ovarian cancer; favorable response rates in a phase I/II study are associated with an immunotherapeutic effect. Gynecol Oncol. 2020 Jun;157(3):578-584. doi: 10.1016/j.ygyno.2020.02.034. Epub 2020 Apr 5. PMID 32265057